CLINICAL TRIAL: NCT03813290
Title: A Neuro-Technological Intervention for Adolescents With Generalised Anxiety Disorder (GAD): A Feasibility Trial
Brief Title: A Neuro-Technological Intervention for Adolescents With GAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore General Hospital (Other); Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Lim Choon Guan, Senior Consultant and Deputy Chief, National Healthcare Group, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DSRB A/2018/00693
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Generalised Anxiety Disorder
Keywords: Brain Computer Interface; Neuro technological intervention; Neurofeedback
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neuro-Technological Intervention (Experimental): Participants will attend a total of 8 x 30 minutes intervention sessions (twice a week) for four consecutive weeks, starting within 1 week after baseline assessment.
  Participants will also be required to fill up some questionnaires at baseline and post-intervention visits.
  Interventions: Device: Neuro-technological Intervention

INTERVENTIONS:
Device: Neuro-technological Intervention — During the intervention sessions, participants will don a head-mounted VR display set and a mobile EEG-biosensor. Each session will begin with a brief audio-guided mindfulness practice, follow by a 15 minutes VR game. Game performances will be influenced by individual's level of anxiety arousal and ability to regulate it.
  Other Names: Brain Computer Interface; Mindfulness based Intervention

SUMMARY:
This study aims to evaluate the safety and acceptability of a basic neuro-technological intervention in the treatment of adolescents with Generalised Anxiety Disorder (GAD). Our technology will deliver a mindfulness-based anxiety regulation intervention through a neuro- / bio-feedback-based virtual reality (VR) game interface that is driven by a novel algorithm.

DETAILED DESCRIPTION:
This study is a single-arm open-label test of feasibility. The recruitment target is 30. Outpatient adolescents diagnosed with GAD will be recruited to undergo 8 x 30 minutes intervention sessions over 4 weeks. Participants who are enrolled will continue to receive treatment-as-usual prescribed by their treating psychiatrist, except for the use of psychotropics. This population is selected as they could elucidate whether our intervention can be beneficial as an early intervention program for GAD.

During the 8 bi-weekly intervention sessions, participants will don a head-mounted VR display set and a mobile EEG-biosensor. The hardwares are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 to 18 years of age inclusive
* Literate in English Language
* Newly diagnosed with Generalised Anxiety Disorder: current episode, based on Computerised Diagnostic Interview Schedule for Children (C-DISC)
* If on medication, dosage stable or unchanged for at least preceding 8 weeks
* Has parental consent

Exclusion Criteria:

* Diagnosis (as defined by DSM-5) of: anxiety disorder induced by medication, substance, or another medical condition; obsessive compulsive disorder; bipolar disorder; any psychotic disorder (lifetime); intellectual disability (i.e. IQ<70); autism spectrum disorder; attention-deficit/hyperactivity disorder
* History of substance or drug use disorder (as per DSM-5 criteria) within the last 3 months
* Neurological disorders or insults (e.g. epilepsy, cerebrovascular accidents)
* Metal in the cranium, skull defects, or skin lesions on scalp (e.g. cuts, abrasion, rash) at proposed electrode sites
* Irregular heart rhythms or heart problems
* Severe visual or hearing impairment
* Prior experience with mindfulness-based therapy (e.g. mindfulness-based stress reduction [MBSR], mindfulness-based cognitive therapy [MBCT])

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Usability Questionnaire | Week 4
  Usability questionnaire measures participants' experience with the neuro-technological intervention devices and software. Subscale with12 items asking about overall comfort and usability are included, with scale range of 1 to 4 (1 - very false for me, 2 - False, 3 - True, 4 - Very true for me). Subsequent 27-items subscale measures participants' experience with the software/virtual reality experience, with scale ranging from 1 to 7 (the lower the rating, the poorer the experience). Total score will be obtained from summing up the scores for each subscale. Higher score means better overall experience with the intervention.

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children (Parent-reported); 2nd Edition | Week 0, 5
  The MASC is a comprehensive, multi-rater assessment of anxiety dimensions in children and adolescents aged 8 to 19 years old. The MASC includes subscales scores for separation anxiety/phobias, GAD index, social anxiety, obsessions & compulsions, physical symptoms and harm avoidance. Raw scores from these subscales will be summed up to obtain the total score. Scale ranges from 0 to 3 (0 - Never, 1 - Rarely, 2 - Sometimes, 3 - Often). Higher raw scores indicate higher anxiety symptoms.
Multidimensional Anxiety Scale for Children (Adolescent-reported); 2nd Edition | Week 0, 5
  The MASC is a comprehensive, multi-rater assessment of anxiety dimensions in children and adolescents aged 8 to 19 years old. The MASC includes subscales scores for separation anxiety/phobias, GAD index, social anxiety, obsessions & compulsions, physical symptoms and harm avoidance. Raw scores from these subscales will be summed up to obtain the total score. Scale ranges from 0 to 3 (0 - Never, 1 - Rarely, 2 - Sometimes, 3 - Often). Higher raw scores indicate higher anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lim Choon Guan, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Child Guidance Clinic, Singapore, Singapore, Singapore